CLINICAL TRIAL: NCT04791436
Title: Oral and Olfactory Complications of Recovered COVID-19 Patients: A Prospective Cohort Study
Brief Title: Oral and Olfactory Complications of Recovered COVID-19 Patients
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Masaryk University (Other); University of Kiel (Other)
Responsible Party: Principal Investigator, Sameh Attia, Head of the Dental Polyclinic, University of Giessen
Other Study IDs: OORCV
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Oral Complication; Dysgeusia; Olfactory Disorder
Keywords: COVID-19; Oral Manifestations; Olfactory Manifestations
MeSH Terms: conditions — Dysgeusia; COVID-19; Oral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Illness: Recovered COVID-19 patients who experienced a mild clinical course
  Interventions: Diagnostic Test: Gustatory and olfactory function test; Diagnostic Test: Molecular assessment of saliva
- Moderate Illness: Recovered COVID-19 patients who experienced a moderate clinical course
  Interventions: Diagnostic Test: Gustatory and olfactory function test; Diagnostic Test: Molecular assessment of saliva
- Severe Illness: Recovered COVID-19 patients who experienced a severe clinical course
  Interventions: Diagnostic Test: Gustatory and olfactory function test; Diagnostic Test: Molecular assessment of saliva

INTERVENTIONS:
Diagnostic Test: Gustatory and olfactory function test — The gustatory and olfactory function will be tested by using the combined Burghart Screening 12 test containing smelling sticks and taste strips (Fa. MediSense, Groningen, Netherlands). Evaluation of taste and smell is performed by offering the sticks/strips and demand a forced multiple choice.
Diagnostic Test: Molecular assessment of saliva — Saliva samples will be taken for molecular biological determination of the oral microbiome. The microbiome is determined at the Institute for Medical Microbiology by 16s-rRNA gene analysis with Next Generation Sequencing and bioinformatics.

SUMMARY:
This cohort study aims to investigate the long-standing chemosensory disorders and oral manifestation after recovery of the COVID-19 illness. A correlation between the long-standing symptoms and the COVID-19 severity grade will be very important to understand and clarify the aetiology of these symptoms.

DETAILED DESCRIPTION:
This prospective cohort study aims to investigate the long-standing chemosensory disorders and oral manifestation after recovery of the COVID-19 illness. A correlation between the long-standing symptoms and the COVID-19 severity grade will be very important to understand and clarify the aetiology of these symptoms.

Study objectives:

1. To describe the frequency and severity of oral signs and chemosensory disorders that persist after the recovery of COVID-19 and to examine whether "taste disorders" can be discriminated into an- or hypogeusia and an- or hyposmia.
2. To report any correlation between the severity grade of COVID-19 and the resulting standing symptoms.
3. To describe the oral microbiome after infection with COVID-19 and to describe possible changes in comparison to normal healthy individuals.

Clinical and -if indicated- radiological examination to assess the long-term oral and chemosensory impairment and complaints of COVID-19 patients after their recovery shall be performed in an interdisciplinary setting of Maxillofacial Surgery, ENT and Medical Microbiology.

The study subjects will be divided into three groups according to the severity grade of illness: non-hospitalized, hospitalized, and intensive care patients. All adult COVID-19 recovery patients (exceeding the age of 18) will be included in the study. The time between illness and study recruitment shall be at least 3 months. Exclusion criteria are psychiatric or neurological diseases, previous trauma, surgery or radiotherapy in the oral or nasal cavities, pre-existing taste or smell dysfunctions or chronic rhinosinusitis.

The study variables include age, sex, co-morbidities, possible causes of exclusion from the study. The oral health assessment will be performed by examination of: periodontal status, assessment of oral lesions, a radiological examination by using panoramic x-ray if clinically indicated, photo documentation, objective evaluation of the olfactory and gustatory functions with psychophysical tests. The gustatory and olfactory function will be tested by using the combined Burghart Screening 12 test containing smelling sticks and taste strips (Fa. MediSense, Groningen, Netherlands). Evaluation of taste and smell is performed by offering the sticks/strips and demand a forced multiple choice.

ELIGIBILITY:
Inclusion Criteria:

* All adult COVID-19 recovery patients (exceeding the age of 18) will be included in the study. The time between illness and study recruitment shall be at least 3 months.

Exclusion Criteria:

* Exclusion criteria are psychiatric or neurological diseases, previous trauma, surgery or radiotherapy in the oral or nasal cavities, pre-existing taste or smell dysfunctions or chronic rhinosinusitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be divided into three groups according to the severity grade of illness: non-hospitalized, hospitalized, and intensive care patients.
Sampling Method: Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
Periodontal health | At least 3 months after recovery of COVID-19
  Community Periodontal Index (CPI) of the World Health Organization (WHO) will be used to assess periodontal health (continuous variable)
Oral mucocutaneous lesions | At least 3 months after recovery of COVID-19
  An intraoral examination will be carried out to assess the presence of any mucocutaneous lesions (dichotomous variable)
Gustatory function | At least 3 months after recovery of COVID-19
  Burghart Sniffin' Sticks "Screening 12 Test" will be used to assess gustatory function (continuous variable)
Olfactory function | At least 3 months after recovery of COVID-19
  Burghart Sniffin' Sticks "Screening 12 Test" will be used to assess olfactory function (continuous variable)

CONTACTS AND LOCATIONS:
Locations (1):
- Justus-Liebig University, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attia S, Howaldt HP. Impact of COVID-19 on the Dental Community: Part I before Vaccine (BV). J Clin Med. 2021 Jan 14;10(2):288. doi: 10.3390/jcm10020288. PMID 33466777
- [Background] Bottger S, Zechel-Gran S, Streckbein P, Knitschke M, Hain T, Weigel M, Wilbrand JF, Domann E, Howaldt HP, Attia S. A New Type of Chronic Wound Infection after Wisdom Tooth Extraction: A Diagnostic Approach with 16S-rRNA Gene Analysis, Next-Generation Sequencing, and Bioinformatics. Pathogens. 2020 Sep 28;9(10):798. doi: 10.3390/pathogens9100798. PMID 32998201
- [Background] Ammar N, Aly NM, Folayan MO, Mohebbi SZ, Attia S, Howaldt HP, Boettger S, Khader Y, Maharani DA, Rahardjo A, Khan I, Madi M, Shamala A, Al-Batayneh OB, Rashwan M, Pavlic V, Cicmil S, Galluccio G, Polimeni A, Mancino D, Arheiam A, Dama MA, Nyan M, Phantumvanit P, Kim JB, Choi YH, Castillo JL, Joury E, Abdelsalam MM, Alkeshan MM, Hussein I, Vukovic AP, Iandolo A, Kemoli AM, El Tantawi M. Knowledge of dental academics about the COVID-19 pandemic: a multi-country online survey. BMC Med Educ. 2020 Nov 2;20(1):399. doi: 10.1186/s12909-020-02308-w. PMID 33138810
- [Background] Ammar N, Aly NM, Folayan MO, Khader Y, Virtanen JI, Al-Batayneh OB, Mohebbi SZ, Attia S, Howaldt HP, Boettger S, Maharani DA, Rahardjo A, Khan I, Madi M, Rashwan M, Pavlic V, Cicmil S, Choi YH, Joury E, Castillo JL, Noritake K, Shamala A, Galluccio G, Polimeni A, Phantumvanit P, Mancino D, Kim JB, Abdelsalam MM, Arheiam A, Dama MA, Nyan M, Hussein I, Alkeshan MM, Vukovic AP, Iandolo A, Kemoli AM, El Tantawi M. Behavior change due to COVID-19 among dental academics-The theory of planned behavior: Stresses, worries, training, and pandemic severity. PLoS One. 2020 Sep 29;15(9):e0239961. doi: 10.1371/journal.pone.0239961. eCollection 2020. PMID 32991611